CLINICAL TRIAL: NCT00755066
Title: The Effect of Intranasal Corticosteroid on the Immune Response Following Nasal Allergen Challenge in Patients Suffering From Seasonal Allergic Rhinitis
Brief Title: Effect of Intranasal Corticosteroids on Systemic Allergen Specific IgE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Allergy Centre Vienna West (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2505; EudraCT 2005-004274-24
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- F (Experimental): Fluticasone propionate 200 µg intranasal
  Interventions: Drug: Fluticasone propionate
- P (Placebo Comparator): Placebo intranasal spray
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone propionate — 200 µg intranasal, 4 weeks, od.
  Arms: F
Drug: Placebo — Placebo intranasal spray
  Arms: P

SUMMARY:
Evaluation of the effect of fluticasone propionate vs placebo applied as nasal spray on the increase of allergen-specific serum IgE levels following nasal exposure to recombinant allergens. Nasal sprays will be applied for four weeks starting two weeks before nasal provocation and serum IgE levels will be followed during eight weeks after nasal provocation.

ELIGIBILITY:
Inclusion Criteria:

* male or female 18-50 years of age
* moderate to severe allergic rhinitis to grass and/or birch pollen for at least two seasons according to history
* sensitization to rPhl p 5 and rBet v 1 as demonstrated by UniCAP within a range from 3.0-80 kUA/l and a positive (wheal diameter >= 3 mm larger than the negative control and half of the histamine control) SPT with rPhl p 5 and rBet v 1 at 20 µg/ml
* willingness to comply with the study protocol
* written informed consent

Exclusion Criteria:

* perennial allergic rhinitis
* history of asthma necessitating treatment
* FEV1 <70% of predicted value
* abnormalities at auscultation of heart or lungs
* history of anaphylaxis
* severe atopic dermatitis
* total serum IgE >2000 kU/l
* previous or ongoing immunotherapy (subcutaneous or sublingual) to grass or birch pollen
* nasal provocation testing during the previous six month
* known allergy/intolerance to fluticasone propionate or loratadine
* known allergy/intolerance to cellulose, polysorbate, phenylethyl alcohol, benzalkonium chloride
* contraindications for the use of INCS:
* acute or chronic infections of the upper respiratory tract
* surgery of the nose during the previous year
* hypersensitivity to components of the drug
* contraindications for nasal provocation test
* acute rhinosinusitis
* acute allergic reaction of the immediate type at other organs
* nasal polyposis or significant nasal anatomical deformities
* vasomotor rhinitis
* autoimmune disease, chronic or acute infectious disease, malignancy
* severe psychological disorder
* treatment with systemic or topical (intranasal, inhaled, external) corticosteroids from 3 month prior to the study
* treatment with other immunosuppressant drugs from 6 month prior to the study
* treatment with antihistamines or disodium cromoglycate from 2 weeks prior to the study
* treatment with intranasal adrenergic drugs from 3 days prior to the study
* treatment with systemic adrenergic drugs
* treatment with psychopharmacological drugs from 2 weeks prior to the study
* cardiovascular or pulmonary disease
* contraindication for adrenaline
* participation in any other clinical trial within the previous 3 month
* pregnant, lactating or sexually active women with childbearing potential who are not using a medically accepted birth control method
* a mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude
* known alcohol or drug addiction or abuse
* unlikelihood to be able to complete the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)

PRIMARY OUTCOMES:
Allergen specific IgE levels | 8 weeks

SECONDARY OUTCOMES:
Allergen specific IgG 1-4, IgM, IgA levels | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Horak, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Allergy Centre Vienna West, Vienna, Austria

REFERENCES:
- [Derived] Egger C, Lupinek C, Ristl R, Lemell P, Horak F, Zieglmayer P, Spitzauer S, Valenta R, Niederberger V. Effects of nasal corticosteroids on boosts of systemic allergen-specific IgE production induced by nasal allergen exposure. PLoS One. 2015 Feb 23;10(2):e0114991. doi: 10.1371/journal.pone.0114991. eCollection 2015. PMID 25705889